CLINICAL TRIAL: NCT03984435
Title: A Qualitative Study Exploring Patient Experiences of Comfort During Radiotherapy and Radiographer Views of Managing Patient Comfort During the Delivery of Radiotherapy
Brief Title: Patients' and Radiographers' Experiences and Views of Comfort Management in Radiotherapy
Acronym: COMFORT
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of the West of England (Other)
Collaborators: Somerset NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: HAS.19.02.126
Record Dates: First submitted 2019-06-10; First posted 2019-06-13 (Actual); Last update posted 2019-06-13 (Actual); Status verified 2019-06

CONDITIONS: Cancer
Keywords: Radiotherapy; Experiences; Comfort management; Patients; Radiographers
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients: Patients with a diagnosed malignancy who have been referred for radiotherapy with extended treatment time (>10 minutes)
- Radiographers: Radiographers from radiotherapy departments in the UK who deliver radiotherapy

SUMMARY:
A qualitative study exploring patient experiences of comfort during radiotherapy and radiographers' views of managing patient comfort during the delivery of radiotherapy

DETAILED DESCRIPTION:
Patients undergoing radiotherapy treatment for cancer frequently express their feelings of discomfort during the procedure, especially those who require radiotherapy with extended treatment times. This problem was explored by informal questioning of patients who revealed that this is a problem and causes distress and discomfort but that it was being accepted as being part of the treatment. In healthcare, several interventions have been used to improve the comfort of patients. In radiotherapy, there have been examples where positioning or relaxation has improved the patient's comfort. Literature searches have revealed some comfort interventions that can be used during radiotherapy treatment which may be possible interventions.

With the consent of the patient, it is intended to establish the patients' experience and views of comfort and comfort management during radiotherapy. Radiographers' experiences and views of managing patient comfort during radiotherapy will also be explored. It will also be essential to explore what would be the most ideal solution to comfort management, or how comfort could be improved, from the perspective of both patients and radiographers.

ELIGIBILITY:
Inclusion Criteria:

Patients:

1. diagnosed with a malignancy;
2. aged over 18 years owing to different treatment options for children and young adults;
3. recently referred for radiotherapy, currently receiving treatment or had had radiotherapy within the previous 3 months;
4. treatment delivery time exceeding 10 minutes (the time the patient is immobilised on the radiotherapy couch).

Therapeutic radiographers:

1. practicing Therapeutic radiographers;
2. administering radiotherapy with treatment delivery times exceeding 10 minutes per radiotherapy treatment session (the time the patient is immobilised on the radiotherapy couch).

Exclusion Criteria:

Patients:

1. patients with treatment delivery time below 10 minutes;
2. unable to communicate in English.

Therapeutic Radiographers:

1. student Therapeutic radiographers,
2. no more than two radiographers from the same radiotherapy department.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients: any person receiving radiotherapy at Musgrove Park Hospital, Taunton, with Therapeutic radiographers: no more than two from any radiotherapy department throughout the UK.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2019-02-08 (Actual); Primary Completion 2019-08-15 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
Experiences of comfort during radiotherapy - qualitative (non-standard outcome measure) | Duration of radiotherapy and up to three months after
  This is qualitative research and the outcomes are derived from transcribed interviews analysed thematically generating codes, themes and sub-themes of patient and radiographers lived experiences of comfort during radiotherapy.

CONTACTS AND LOCATIONS:
Overall Officials: Simon D Goldsworthy, MSc, Principal Investigator — Principal Research Radiographer
Locations (1):
- Musgrove Park Hospital, Taunton, Somerset, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Access to anonymised interview transcripts on written request to UWE Bristol
Supporting Information: Study Protocol, CSR
Time Frame: 10 years from production of data
Access Criteria: Via DMPonline
URL: http://dmponline.dcc.sc.uk

REFERENCES:
- [Background] Schnur JB, Ouellette SC, Bovbjerg DH, Montgomery GH. Breast cancer patients' experience of external-beam radiotherapy. Qual Health Res. 2009 May;19(5):668-76. doi: 10.1177/1049732309334097. PMID 19380502
- [Background] Arcangeli S, Scorsetti M, Alongi F. Will SBRT replace conventional radiotherapy in patients with low-intermediate risk prostate cancer? A review. Crit Rev Oncol Hematol. 2012 Oct;84(1):101-8. doi: 10.1016/j.critrevonc.2011.11.009. Epub 2012 Jan 17. PMID 22257653
- [Background] Gestaut MM, Thawani N, Kim S, Gutti VR, Jhavar S, Deb N, Morrow A, Ward RA, Huang JH, Patel M. Single fraction spine stereotactic ablative body radiotherapy with volumetric modulated arc therapy. J Neurooncol. 2017 May;133(1):165-172. doi: 10.1007/s11060-017-2428-6. Epub 2017 Apr 13. PMID 28409420
- [Background] Chang JH, Gandhidasan S, Finnigan R, Whalley D, Nair R, Herschtal A, Eade T, Kneebone A, Ruben J, Foote M, Siva S. Stereotactic Ablative Body Radiotherapy for the Treatment of Spinal Oligometastases. Clin Oncol (R Coll Radiol). 2017 Jul;29(7):e119-e125. doi: 10.1016/j.clon.2017.02.004. Epub 2017 Feb 23. PMID 28237218
- [Background] Dawson LA, Balter JM. Interventions to reduce organ motion effects in radiation delivery. Semin Radiat Oncol. 2004 Jan;14(1):76-80. doi: 10.1053/j.semradonc.2003.10.010. PMID 14752735
- [Background] Cheng. F, Wang.W. Factors influencing comfort level in head and neck neoplasm patients receiving radiotherapy. Int J Nur Scie. 2014; 1 (4): 394-399
- [Background] Cox.J. Davison.A. Comfort as a determiner of treatment position in radiotherapy of the male pelvis. Radiog. 2005; 11 (2): 109-115
- [Background] Goldsworthy.SD, Tuke.K, Latour.J.M. A focus group consultation round exploring patient experiences of comfort during radiotherapy for head and neck cancer; Journal of Radiotherapy in Practice; 2016; 15 (2)143-149
- [Background] Pineau,C. The psychological meaning of comfort. International Review of Applied Psychology. 1982. Vol 31, 271-283
- [Background] Kolcaba K, Steiner R. Empirical evidence for the nature of holistic comfort. J Holist Nurs. 2000 Mar;18(1):46-62. doi: 10.1177/089801010001800106. PMID 11847691
- [Background] Kolcaba K, Tilton C, Drouin C. Comfort Theory: a unifying framework to enhance the practice environment. J Nurs Adm. 2006 Nov;36(11):538-44. doi: 10.1097/00005110-200611000-00010. PMID 17099440
- [Background] Braun V. Clarke V. Using thematic analysis in psychology. Qualitative Research in Psychology; 2006 July 3: 77-101
- [Background] Carter N, Bryant-Lukosius D, DiCenso A, Blythe J, Neville AJ. The use of triangulation in qualitative research. Oncol Nurs Forum. 2014 Sep;41(5):545-7. doi: 10.1188/14.ONF.545-547. PMID 25158659
- [Derived] Goldsworthy S, Latour JM, Palmer S, McNair HA, Cramp M. A thematic exploration of patient and radiation therapist solutions to improve comfort during radiotherapy: A qualitative study. J Med Imaging Radiat Sci. 2023 Dec;54(4):603-610. doi: 10.1016/j.jmir.2023.07.008. Epub 2023 Jul 20. PMID 37479627
- See also: COMFORT study Twitter account — https://twitter.com/ComfortStudy